CLINICAL TRIAL: NCT01511289
Title: A Phase 3 Multinational, Multi-center, Open-Label, Randomized Study of the Efficacy of Radotinib Versus Imatinib in Newly Diagnosed Ph+ CML Patients in Early Chronic Phase
Brief Title: Radotinib Versus Imatinib in Newly Diagnosed Philadelphia Chromosome and Chronic Myeloid Leukemia Chronic Phase Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IY5511A3001
Record Dates: First submitted 2012-01-03; First posted 2012-01-18 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome; Bone Marrow Diseases; Hematologic Diseases
Keywords: Radotinib; CML-CP; Chronic Myeloid Leukemia, chronic phase
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome; Bone Marrow Diseases; Hematologic Diseases; Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate; 4-methyl-N-(3-(4-methylimidazol-1-yl)-5-trifluoromethylphenyl)-3-(4-pyrazin-2-ylpyrimidin-2-ylamino)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Imatinib (Active Comparator): Imatinib 400mg QD
  Interventions: Drug: Imatinib
- Radotinib 600mg (Experimental): Radotinib 300mg BID
  Interventions: Drug: Radotinib
- Radotinib 800mg (Experimental): Radotinib 400mg BID
  Interventions: Drug: Radotinib

INTERVENTIONS:
Drug: Imatinib — 400mg/Tab, QD
  Other Names: Glivec; Gleevec
  Arms: Imatinib
Drug: Radotinib — 100mg or 200mg/Capsule, 300mg or 400mg BID
  Other Names: IY5511HCl
  Arms: Radotinib 600mg; Radotinib 800mg

SUMMARY:
In this study, the efficacy and safety of two radotinib doses, 300 mg twice daily and 400 mg twice daily, will be compared with imatinib 400 mg once daily in newly diagnosed patients with Philadelphia chromosome-positive (Ph+) Chronic Myelogenous Leukemia in the chronic phase (CML-CP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of chronic phase CML within last 3 months
* Patients with cytogenetically confirmed Ph positive CML in early chronic phase

Exclusion Criteria:

* Patients with Philadelphia chromosome negative but BCR-ABL positive CML
* Patients who used imatinib for 8 days or longer before study entry
* Patients who had been treated with other targeted anti-cancer therapy, except for Hydrea or Agrylin, which inhibits the growth of leukemic cells
* Patients with impaired cardiac function
* Cytologically confirmed CNS involvement
* Severe or uncontrolled chronic medical condition
* Other significant congenital or acquired bleeding disorders that are not related to underlying leukemia
* Patients who had a major surgery within 4 weeks prior to study entry or has not recovered from side effects of such surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2011-08; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Rate of Major Molecular Response(MMR) by 12 months | 12 months
  Rate of Major Molecular Response (MMR) at Any Time within 12 months. MMR by 12 months will be assessed as responder if the patient has response at any time within 12 months.
  A major molecular response rate is defined as the ratio (%) of BCR-ABL/ABL ≤ 0.1% by international scale or a 3-log reduction in BCR-ABL transcript level from standardized baseline, as measured by standardized RQ-PCR assay.

SECONDARY OUTCOMES:
Rate of complete cytogenetic response (CCyR) by 12 months | 12 months
  Complete cytogenetic response is defined as complete disappearance of Philadelphia-positive in at least 20 metaphases examined. Chromosome analysis performed on less than 20 metaphases will not be accepted for this study
Rate of complete molecular response (CMR) by 12 months | 12 months
  Complete molecular response is defined as negative BCR-ABL transcript levels, as measured twice by the internationally standardized RQ-PCR assay.
  The rate of complete molecular response by cycle 12 is defined as an at least 4.5 log reduction in BCR-ABL transcript levels from standardized baseline or BCR-ABL/ABL % ≤ 0.005% by the international scale.
Rate of major molecular response (MMR) at 12 months | 12 month
  Rate of Major Molecular response will be assessed at 12 months at that timepoint.
  Number of Participants With Major Molecular Response (MMR) at 12 months.
Rate of subjects with disease progression | 12 months
  Disease progression by month 12 will be compared between each groups.

CONTACTS AND LOCATIONS:
Overall Officials: IL-YANG PHARM, Study Director — IL-YANG Pharmaceutical. Co., LTD
Locations (14):
- Local Institution, Jakarta, Indonesia
- Philippines (2):
  - Local Institution, Batangas
  - Local Institution, Manila
- South Korea (10):
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Gyeonggi-do
  - Local Institution, Incheon
  - Local Institution, Jeollabuk-do
  - Local Institution, Jeonnam
  - Local Institution, Seoul
  - Local Institution, Ulsan
  - Local Institution, Wŏnju
- Local Institution, Bangkok, Thailand

REFERENCES:
- [Derived] Kwak JY, Kim SH, Oh SJ, Zang DY, Kim H, Kim JA, Do YR, Kim HJ, Park JS, Choi CW, Lee WS, Mun YC, Kong JH, Chung JS, Shin HJ, Kim DY, Park J, Jung CW, Bunworasate U, Comia NS, Jootar S, Reksodiputro AH, Caguioa PB, Lee SE, Kim DW. Phase III Clinical Trial (RERISE study) Results of Efficacy and Safety of Radotinib Compared with Imatinib in Newly Diagnosed Chronic Phase Chronic Myeloid Leukemia. Clin Cancer Res. 2017 Dec 1;23(23):7180-7188. doi: 10.1158/1078-0432.CCR-17-0957. Epub 2017 Sep 22. PMID 28939746